CLINICAL TRIAL: NCT06248268
Title: Differences Between Suicide Attempters and Suicide Ideators. Influence of the Brief Therapy ASSIP on Neuropsychological Correlates and Psychological Process Factors (NePsyASSIP HT) - Project 1
Brief Title: Neuropsychological Patterns of Suicide Ideators and Suicide Attempters
Acronym: NePsyAssip HT
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02504 (Project 1)
Record Dates: First submitted 2023-03-13; First posted 2024-02-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inhibitory Control; Locus of Control; Self Efficacy; Suicide, Attempted; Suicidal Ideation; Attention
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Suicide attempters: Patients with at least one previous suicide attempt
  Interventions: Other: (Neuro-)psychological assessment
- Suicide ideators: Patients with suicidal thoughts, but no previous suicide attempt
  Interventions: Other: (Neuro-)psychological assessment
- Clinical control group: Patients without suicidal behavior and thoughts
  Interventions: Other: (Neuro-)psychological assessment
- Healthy controls: Healthy persons without suicidal behavior and thoughts
  Interventions: Other: (Neuro-)psychological assessment

INTERVENTIONS:
Other: (Neuro-)psychological assessment — The measurement, which takes place 1 week after the informed consent, aims to determine the distinct (neuro-) psychological patterns of suicidal behavior versus suicidal ideation, in comparison to two control groups.

SUMMARY:
The present study consists of 3 projects in total and aims to investigate the (neuro-) psychological patterns from suicidal ideation to suicidal behavior as well as the effects and feasibility of ASSIP Home Treatment.

The overall aim of project 1 is to determine (neuro-) psychological differences between suicide attempters, suicide ideators, a clinical control group, and healthy controls. Study participants in project 1 will participate in a one-time (neuro-) psychological assessment.

Project 1 of this study is an observational cross-sectional study with four groups that will be conducted at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland): Patients with at least one suicide attempt in their past (SUAT), patients with suicidal ideation (SUID), patients from the same clinical cohort, without neither suicidal behavior or ideation (CLIN) and the healthy group (HLTH). The cohorts to be examined (SUAT & SUID) will be compared to the two control groups (CLIN & HLTH). Only people who have signed the informed consent and meet the eligibility criteria can participate in this study.

DETAILED DESCRIPTION:
Purpose and aims:

The present study consists of 3 projects in total and aims to investigate the (neuro-) psychological patterns from suicidal ideation to suicidal behavior as well as the effects and feasibility of ASSIP Home Treatment.

The aim of this project is to distinguish the (neuro-) psychological patterns of suicide ideators from suicide attempters by investigating four experimental groups. For this purpose, neuropsychological functioning, as well as psychological process factors, are analyzed. Patients with at least one prior suicide attempt are compared to patients with suicidal ideation, to a clinical control group, as well as to healthy controls. For this project, patients who are being treated at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland) at the time of the project will be requested. Afterwards, participants with a suicide attempt in their history will also be asked to participate in the longitudinal part of the study, which is Project 2.

Background:

In Switzerland, approximately three people die by suicide every day, and suicide attempts exceed this number by far. As a previous suicide attempt is one of the strongest predictors of a completed suicide, it is of utmost importance to identify the people at risk. However, research has shown that traditional risk factors (e.g., depression, psychiatric disorder, etc.) reliably predict suicidal ideation but poorly predict suicidal behavior. Furthermore, while effective suicide-specific interventions exist, up to 50% of the suicide attempters reject the recommended treatment, and around 60% discontinue treatment after one session. Hence, a different approach is required. In this study, three projects will be conducted. In Project 1, (neuro-) psychological patterns of suicide attempters will be identified by comparing the following four different groups:

1. patients with a prior suicide attempt (SUAT),
2. patients with no prior suicide attempt but suicidal ideation (SUID),
3. a general patient group (CLIN), and
4. a healthy control group (HLTH).

Project 2 will investigate how these patterns are modulated by the efficacious brief therapy ASSIP. In Project 3, the feasibility, effects and cost-effectiveness of the ASSIP Home Treatment will be investigated.

Study design of Project 1:

Project 1 of this study is a quantitative cross-sectional and observational study with four groups that will be conducted at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland): Patients with at least one suicide attempt in their past (SUAT), patients with suicidal ideation (SUID), patients from the same clinical cohort without suicidal behavior or ideation (CLIN), and the healthy group (HLTH). The cohorts to be examined (SUAT & SUID) will be compared to two control groups (CLIN & HLTH). Study participants in Project 1 will participate in a one-time (neuro-) psychological assessment. To account for the heterogeneity in suicide attempters, suicide ideators, generally clinical patients and healthy controls, the samples will be balanced for age, gender and treatment setting by group matching.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling the following inclusion criteria are eligible for the study:

* Informed consent as documented by signature
* Age ≥ 18 years

Additional inclusion criterion for the SUAT group in project 1:

• At least one previous suicide attempt

Additional inclusion criterion for the SUID group in project 1:

• Suicidal ideation

Additional inclusion criterion for the CLIN group in project 1:

• Current psychiatric disorder treated on an inpatient, day-care or outpatient basis For the HLTH group, no further inclusion criteria are formulated.

Exclusion Criteria:

The presence of any one of the following exclusion criteria leads to exclusion of the subject:

* Serious cognitive impairment
* Any current psychotic disorder
* Any current medication, which substantially impairs the attention span, reaction rate or any other relevant cognitive functions
* Inability to follow the procedures of the study (e.g., insufficient mastery of the German language, previous enrolment into the current study)

Additional exclusion criterion for the SUID group:

• Previous suicidal behavior

Additional exclusion criteria for the CLIN and HLTH groups:

* Previous suicidal behavior
* Suicidal ideation

Additional exclusion criterion for the HLTH group:

• Current psychiatric disorder treated on an inpatient, day-care or outpatient basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This quantitative cross-sectional study with four groups will be conducted at the University Hospital of Psychiatry and Psychotherapy, Bern. Patients with at least one suicide attempt in their past (SUAT), patients with suicidal ideation (SUID), patients from the same clinical cohort without neither suicidal behavior or ideation (CLIN), and the healthy group (HLTH). The cohorts to be examined (SUAT & SUID) will be compared to two control groups (CLIN & HLTH).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in Inhibitory Control | The assessment takes place 1 day to 1 week after informed consent.
  The Go/No-Go task is a cognitive task to assess an individual's ability to inhibit a prepotent response. It is used to measure impulse control and response inhibition. The task requires participants to respond ("Go" response) to one type of stimulus and to withhold or inhibit their response ("No-Go" response) to another type of stimulus. The Go/No-Go task yields measures such as reaction time, accuracy, and the ability to inhibit responses. Reaction times can vary widely, and accuracy is often expressed as a percentage of correct responses. Lower reaction times and higher accuracy in withholding responses (No-Go trials) indicate better inhibitory control and cognitive performance.

SECONDARY OUTCOMES:
Selective Attention and Interference Control | The assessment takes place 1 day to 1 week after informed consent.
  The Stroop task is a cognitive psychology test that evaluates an individual's ability to selectively attend to information while inhibiting interference from irrelevant stimuli. The Stroop task measures the time taken to complete tasks and the accuracy of responses. The primary measures are the time taken to complete the task and the number of errors. Lower completion times and fewer errors indicate better cognitive control and attentional focus. Lower scores (faster completion times and fewer errors) are associated with better outcomes, reflecting more efficient cognitive processing and interference control. Higher scores, if used to quantify errors or time taken, are associated with a worse outcome, indicating greater interference and potentially reduced cognitive control.

OTHER OUTCOMES:
Mental abilities like attention, working memory and visuomotor speed as well as mental flexibility | The assessment takes place 1 day to 1 week after informed consent.
  The Trail Making Test (TMT-A/B) is a neuropsychological test that assesses visual attention and task-switching abilities. It consists of two parts (Part A and Part B) and measures the time taken to complete each part. The score is typically represented as the time (in seconds) taken to complete the task. Lower scores (faster completion times) are generally considered better outcomes, indicating more efficient visual attention, processing speed, and cognitive flexibility. Higher scores (longer completion times) may suggest difficulties in these cognitive domains and are typically associated with worse outcomes.
Attention and Concentration Abilities | The assessment takes place 1 day to 1 week after informed consent.
  The D2 Test of Attention and Concentration is a neuropsychological test used to assess selective and sustained attention. It is employed to evaluate an individual's visual scanning, concentration, and information processing speed. The D2 Test involves scoring based on the number of correctly marked items minus the number of errors. The scoring method considers both the quantity and accuracy of responses. The goal is to mark as many target items as possible within a specified time limit while avoiding errors. A higher score is considered a better outcome, indicating more correct responses and effective attention and concentration.
Sociodemographic data | The assessment takes place 1 day to 1 week after informed consent.
  The Sociodemographic Questionnaire (DEMO) is a 30-item questionnaire that was developed to collect sociodemographic (e.g., gender, socioeconomic status, professional status, relationship satisfaction) and health-related data (e.g., medication, inpatient and outpatient treatment).
Diagnostic and Statistical Manual 5 (DSM-V) and International Classification of Diseases 10 (ICD-10) psychiatric disorders | The assessment takes place 1 day to 1 week after informed consent.
  The Mini-DIPS is a short, structured clinical interview for diagnosing mental disorders and is based on the DIPS-OA. The Mini-DIPS allows for a quick yet reliable diagnosis. It is applicable in adulthood and captures lifetime diagnoses, current and past diagnoses, based on the criteria of DSM-5 and ICD-10. The Mini-DIPS covers the mental disorders most commonly observed in clinical settings.
Suicidal Ideation | The assessment takes place 1 day to 1 week after informed consent.
  The Beck Scale for Suicide Ideation (BSS) is a clinical assessment tool designed to measure the severity of suicidal ideation in individuals. It is used in clinical and research settings to assess the risk of suicide. The BSS consists of 19 items, and each item is scored on a 3-point scale (0 to 2). The total score, which ranges from 0 to 38, reflects the severity of suicidal ideation. The minimum score is 0, indicating no suicidal ideation and the maximum score is 38, indicating the highest level of suicidal ideation. Higher scores indicate a greater severity of suicidal ideation, and thus, higher scores are generally associated with a worse outcome.
Depressive Symptoms | The assessment takes place 1 day to 1 week after informed consent.
  The Beck Depression Inventory (BDI-II) is a self-assessment questionnaire and contains 21 items which assess the severity of depressive symptoms. A participant's score is calculated by summing up the scores from each item. The total score ranges from 0 to 63. Values between 0 and 11 lie within the norm, between 11 and 17 moderate depressive symptoms and a total score up to 18 is assessed as a clinically relevant depressive disorder.
Psychological Pain | The assessment takes place 1 day to 1 week after informed consent.
  The Mee-Bunney Psychological Pain Assessment Scale (MBPPAS) is a 10-item self-report questionnaire to assess intensity and frequency of psychological pain. Psychological pain is defined as an experience of unbearable agony which can be linked to a psychiatric disorder. Each of the 10 items is rated on a 5-point Likert scale from 1 (never) to 5 (always) or from 1 (none) to 5 (unbearable). The item scores are added up to a total score. A higher score indicates higher psychological pain.
General Sense of Self-Efficacy | The assessment takes place 1 day to 1 week after informed consent.
  The General Self-Efficacy Scale (GSE) is a 10-item self-report questionnaire to assess the general sense of self-efficacy. Items are rated from 1 (do not agree) to 4 (totally agree). A higher score indicates a stronger belief in one's ability to cope with and navigate different situations.
Loneliness | The assessment takes place 1 day to 1 week after informed consent.
  The Three-Item UCLA (University of California, Los Angeles) Loneliness Scale is a short questionnaire with three items from the Revised UCLA Loneliness Scale (R-UCLA). These items can be rated from 1 (hardly ever) to 3 (often). A higher score indicates a higher level of perceived loneliness. The scale is designed to measure subjective feelings of loneliness, so individuals who score higher on the UCLA Loneliness Scale report more frequent experiences of loneliness and social isolation.
Locus of Control | The assessment takes place 1 day to 1 week after informed consent.
  The Internal-External Locus of Control Short Scale-4 (IE-4) is a brief measure designed to assess an individual's locus of control orientation. Locus of control refers to the extent to which individuals believe they control events in their lives. The IE-4 is typically scored by summing the responses to its four items, each rated on a Likert scale. The possible score range is determined by the specific scoring method researchers or practitioners use. The scores may range from 4 to 16, depending on the scoring system employed. Higher scores on the IE-4 may suggest a more internal locus of control, indicating a belief that one has control over their life events. Lower scores may indicate a more external locus of control, suggesting a belief that external factors or luck play a significant role in life events.
Suicide-Related Coping | The assessment takes place 1 day to 1 week after informed consent.
  Coping with suicidal ideation and behavior will be assessed with the Suicide-Related Coping Scale (SRCS). The self-report scale SCRS consists of 17 items, with each rated on a five-point Likert scale from "strongly disagree" = 0 to "strongly agree" = 4. A total SRCS sum score is calculated by inverting the negatively worded items and then summing the 17 items. A higher sum score indicates better suicide-related coping.
Dissociative Experience | The assessment takes place 1 day to 1 week after informed consent.
  The German Dissociation-Tension Scale - 4 (DSS-4) is a four-item brief self-report instrument to assess dissociation. It was developed based on the DSS-acute, a longer scale to measure dissociative symptoms. The four DSS-4 items assess somatic and psychological dissociation and each item is rated on a 10-point Likert scale ranging from "not present" = 0 to "very strong" = 9. Based on the DSS-4, a dissociation score per participant is calculated as the mean of the four items.
Motivational Goals | The assessment takes place 1 day to 1 week after informed consent.
  The Questionnaire for the Analysis of Motivational Schemas (FAMOS) assesses the motivational goals of psychotherapy in terms of central components of motivational schemas in self-report format. The questionnaire FAMOS assesses motivational goals as approach goals on 14 scales and avoidance goals on 9 scales, with a total of 94 items. Each item is rated on a five-point Likert scale. For each scale, the scale mean of the corresponding items is calculated. In addition, three summary values can be calculated: 1) total value for approach goals; 2) total value for avoidance goals; and 3) the ratio of avoidance to approach goals.
Motivational Incongruence | The assessment takes place 1 day to 1 week after informed consent.
  The Incongruence Questionnaire (INK) measures unsatisfactory realization of motivational goals, whereas the personal relevance of motivation is measured in the FAMOS. The questionnaire INK assesses the realization of approach and avoidance goals on 14 and 9 scales, respectively, with a total of 94 items. Each item to assess approach goals is assessed on a five-point Likert scale. For each scale, the mean value of the corresponding item values must be determined. In addition, it is possible to calculate three composite scales: 1) incongruence with avoidance goals; 2) incongruence with approach goals; and 3) total incongruence.
Alcohol Use Screening | The assessment takes place 1 day to 1 week after informed consent.
  The Alcohol Use Disorders Identification Test (AUDIT-C) is an alcohol screen that is used to identify patients who are hazardous drinkers or who may have an active alcohol use disorder. The minimum score (for non-drinkers) is 0, and the maximum possible score is 12. The higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting their health and safety.
Physiologically Experienced Emotional Distress and Arousal | The assessment takes place 1 day to 1 week after informed consent.
  Electrodermal activity (EDA), also known as skin conductance or galvanic skin response, is a valuable physiological marker in suicide research. EDA measures the skin's electrical conductance, reflecting sympathetic nervous system activity. Suicidal individuals often experience heightened emotional distress and arousal, challenging assessment via self-reports alone. EDA offers an objective, non-invasive means to quantify this emotional response, with distinct patterns observed in those at risk of suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Anja C. Gysin-Maillart, PD Dr. phil., Principal Investigator — University of Bern, University Hospital of Psychiatry, Translational Research Center; Lara M. Aschenbrenner, M.Sc., Study Chair — University of Bern, University Hospital of Psychiatry, Translational Research Center
Locations (1):
- University Hospital of Psychiatry and Psychotherapy, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peter, C. and A. Tuch, Suizidgedanken und Suizidversuche in der Schweizer Bevölkerung. Obsan Bulletin. Vol. 7. 2019, Nêuchatel. 2019.
- [Background] Bostwick JM, Pabbati C, Geske JR, McKean AJ. Suicide Attempt as a Risk Factor for Completed Suicide: Even More Lethal Than We Knew. Am J Psychiatry. 2016 Nov 1;173(11):1094-1100. doi: 10.1176/appi.ajp.2016.15070854. Epub 2016 Aug 13. PMID 27523496
- [Background] Ystgaard M, Arensman E, Hawton K, Madge N, van Heeringen K, Hewitt A, de Wilde EJ, De Leo D, Fekete S. Deliberate self-harm in adolescents: comparison between those who receive help following self-harm and those who do not. J Adolesc. 2009 Aug;32(4):875-91. doi: 10.1016/j.adolescence.2008.10.010. Epub 2008 Nov 22. PMID 19028399
- [Background] Klonsky ED, May A. Rethinking impulsivity in suicide. Suicide Life Threat Behav. 2010 Dec;40(6):612-9. doi: 10.1521/suli.2010.40.6.612. PMID 21198330
- [Background] May, A.M. and E.D. Klonsky, What distinguishes suicide attempters from suicide ideators? A meta-analysis of potential factors. Clinical Psychology: Science and Practice, 2016. 23(1): p. 5.
- [Background] Lizardi D, Stanley B. Treatment engagement: a neglected aspect in the psychiatric care of suicidal patients. Psychiatr Serv. 2010 Dec;61(12):1183-91. doi: 10.1176/ps.2010.61.12.1183. PMID 21123401
- [Background] Smith JL, Mattick RP, Jamadar SD, Iredale JM. Deficits in behavioural inhibition in substance abuse and addiction: a meta-analysis. Drug Alcohol Depend. 2014 Dec 1;145:1-33. doi: 10.1016/j.drugalcdep.2014.08.009. Epub 2014 Aug 24. PMID 25195081
- [Background] Nock MK, Park JM, Finn CT, Deliberto TL, Dour HJ, Banaji MR. Measuring the suicidal mind: implicit cognition predicts suicidal behavior. Psychol Sci. 2010 Apr;21(4):511-7. doi: 10.1177/0956797610364762. Epub 2010 Mar 9. PMID 20424092
- [Background] MacLeod CM, MacDonald PA. Interdimensional interference in the Stroop effect: uncovering the cognitive and neural anatomy of attention. Trends Cogn Sci. 2000 Oct 1;4(10):383-391. doi: 10.1016/s1364-6613(00)01530-8. PMID 11025281
- [Background] Reitan, R.M. and D. Wolfson, Category Test and Trail Making Test as measures of frontal lobe functions. The Clinical Neuropsychologist, 1995. 9(1): p. 50-56.
- [Background] Schwarzer, R. and M. Jerusalem, Skala zur allgemeinen Selbstwirksamkeitserwartung. 1999, Berlin: Freie Universität Berlin. 2013.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753
- [Background] Mee S, Bunney BG, Bunney WE, Hetrick W, Potkin SG, Reist C. Assessment of psychological pain in major depressive episodes. J Psychiatr Res. 2011 Nov;45(11):1504-10. doi: 10.1016/j.jpsychires.2011.06.011. Epub 2011 Aug 9. PMID 21831397
- [Background] Hautzinger, M., et al., Beck-depressions-inventar (BDI). Bearbeitung der deutschen Ausgabe. Testhandbuch. Bern: Huber, 1994.
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205